CLINICAL TRIAL: NCT06418165
Title: Vienna Hypothermic Oxygenated Machine Perfusion for Liver Transplantation Study
Brief Title: Vienna Hypothermic Oxygenated Machine Perfusion Study
Acronym: VIHOMPS
Status: Recruiting | Type: Observational
Sponsor: Medical University of Vienna (Other)
Responsible Party: Principal Investigator, David Pereyra, Principal Investigator, Medical University of Vienna
Other Study IDs: 1610/2023
Record Dates: First submitted 2024-05-10; First posted 2024-05-17 (Actual); Last update posted 2024-05-17 (Actual); Status verified 2024-05

CONDITIONS: End Stage Liver Disease; Hepatocellular Carcinoma
Keywords: Liver Transplantation; Hypothermic Oxygenated Machine Perfusion
MeSH Terms: conditions — End Stage Liver Disease; Carcinoma, Hepatocellular

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
In this observational cohort study data on all patients undergoing liver transplantation after hypothermic oxygenated machine perfusion at Medical University of Vienna will be prospectively recorded. Investigation of short- and long-term outcome in this cohort will be conducted.

ELIGIBILITY:
Inclusion Criteria:

* patients undergoing liver transplantation with the use of hypothermic oxygenated machine perfusion
* age ≥ 18 years

Exclusion Criteria:

* pregnancy
* partial grafts
* the anatomical integrity of the liver is not preserved in a way that makes the perfusion of the liver possible

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients listed for and undergoing liver transplantation using a liver graft which was subjected to hypothermic oxygenated machine perfusion
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2018-01-01 (Actual); Primary Completion 2028-12-31 (Estimated); Study Completion 2038-12-31 (Estimated)

PRIMARY OUTCOMES:
Incidence of ischemic-type biliary lesions | Within one year after liver transplantation
  Non-anastomotic stenosis, post-transplant cholangiopathy

SECONDARY OUTCOMES:
Rate of early allograft dysfunction | Evaluated within the first 7 postoperative days
  Deviation of bilirubin, transaminases or international normalised ratio
Rate of primary non-function | Evaluated in the immediate postoperative period, specifically within the first postoperative week
Incidence of re-transplantation | Evaluated in the immediate postoperative period, specifically within the first postoperative week

CONTACTS AND LOCATIONS:
Overall Officials: Gabriela A Berlakovich, Prof, MD, Study Chair — Medical University of Vienna, Division of Transplantation; Georg Györi, MD, Study Director — Medical University of Vienna, Division of Transplantation
Locations (1):
- Medical University of Vienna, Vienna, Austria

IPD SHARING:
Plan to Share IPD: Undecided
data available upon reasonable request and in accordance with appropriate data sharing agreements

REFERENCES:
- [Derived] Pereyra D, Dingfelder J, Riha M, Kacar S, Rauter L, Becker N, Saffarian Zadeh T, Tortopis C, Starlinger P, Ristl R, Silberhumer G, Salat A, Soliman T, Berlakovich G, Gyoeri G. Dual hypothermic oxygenated machine perfusion of the liver reduces post-transplant biliary complications: a retrospective cohort study. Int J Surg. 2024 Dec 1;110(12):7909-7918. doi: 10.1097/JS9.0000000000002115. PMID 39422535